CLINICAL TRIAL: NCT05636657
Title: Comparative Study of Intestinal Color Ultrasound and Capsule Endoscopy in Monitoring Crohn's Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2022-346
Record Dates: First submitted 2022-11-02; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-10

CONDITIONS: Digestive System Disease; Inflammatory Bowel Diseases; Crohn Disease; Crohn Disease of Small Intestine
Keywords: Intestinal Color Ultrasound; Capsule Endoscopy; SUS-CD; CECDAI
MeSH Terms: conditions — Digestive System Diseases; Inflammatory Bowel Diseases; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The disease activity index under intestinal color ultrasound was evaluated by SUS-CD, and the disease activity index under capsule endoscopy was evaluated by CECDAI. All subjects underwent intestinal color ultrasound and capsule endoscopy at baseline and at the third month of treatment. To compare the correlation between SUS-CD and CECDAI before and after treatment, and to compare the role of intestinal color ultrasound and capsule endoscopy in monitoring Crohn's disease in small intestine.

DETAILED DESCRIPTION:
The disease activity index under intestinal color ultrasound was evaluated by SUS-CD, and the disease activity index under capsule endoscopy was evaluated by CECDAI. Active lesions under intestinal color ultrasound were defined as SUS-CD ≥ 1, and active lesions under capsule endoscopy were defined as CECDAI ≥ 3.9. All subjects underwent intestinal color ultrasound and capsule endoscopy at baseline and 3 months after treatment. To compare the correlation between SUS-CD and CECDAI before and after treatment, and to compare the role of intestinal color ultrasound and capsule endoscopy in monitoring Crohn's disease in small intestine.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients diagnosed with Crohn's disease according to the 2019 European Guidelines for Crohn's disease;
* 2.At the time of inclusion, there were active lesions under color ultrasound or capsule endoscopy;
* 3.Voluntarily sign an informed consent form.

Exclusion Criteria:

* 1.Patients with contraindications for capsule endoscopy;
* 2.In the judgment of the investigator, it is not suitable to participate in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with Crohn's disease according to the 2019 European Guidelines for Crohn's disease.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-11-30 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
the Simple Ultrasound Activity Score for Crohn's Disease (SUS-CD) | At baseline
  The Simple Ultrasound Score for Crohn's Disease [SUS-CD] is constituted by Bowel wall thickness (BWT) and colour Doppler. BWT：<3 mm gets 0 score, 3 to 4.9 mm gets 1 score, 5 to 7.9 mm gets 2 scores, and intestinal wall thickness of ≥8 mm gets 3scores. Colour Doppler score：No or single vessel gets 0 score, 2-5 vessels per cm2 gets 1 score, >5 vessels per cm2 gets 2 scores.
the Capsule Endoscopy Crohn's Disease Activity Index(CECDAI) | At baseline
  The CECDAI was designed to evaluate three main parameters of Crohn's disease: inflammation (A), extent of disease (B), and stricture (C), in both the proximal and distal segments of the small bowel. The final score was calculated by adding the two segmental scores: CECDAI =([A1×B1] +C1) +([A2×B2] +C2).
the Simple Ultrasound Activity Score for Crohn's Disease (SUS-CD) | at the third month of treatment
  The Simple Ultrasound Score for Crohn's Disease [SUS-CD] is constituted by Bowel wall thickness (BWT) and colour Doppler. BWT：<3 mm gets 0 score, 3 to 4.9 mm gets 1 score, 5 to 7.9 mm gets 2 scores, and intestinal wall thickness of ≥8 mm gets 3scores. Colour Doppler score：No or single vessel gets 0 score, 2-5 vessels per cm2 gets 1 score, >5 vessels per cm2 gets 2 scores.
the Capsule Endoscopy Crohn's Disease Activity Index(CECDAI) | at the third month of treatment
  The CECDAI was designed to evaluate three main parameters of Crohn's disease: inflammation (A), extent of disease (B), and stricture (C), in both the proximal and distal segments of the small bowel. The final score was calculated by adding the two segmental scores: CECDAI =([A1×B1] +C1) +([A2×B2] +C2).

CONTACTS AND LOCATIONS:
Overall Officials: Xinmei Zhao, doctor, Study Chair — Nanfang Hospital, Southern Medical University
Locations (1):
- NanFang Hospital of Southern Medical University, Guangzhou, Guangdong, China